CLINICAL TRIAL: NCT06191393
Title: Clinical Validation of the Aptitude Medical Systems Metrix COVID/Flu Test for Detection of SARS-CoV-2 and Influenza A/B in Point-of-Care and Non-Laboratory Settings
Brief Title: SARS-CoV-2 and Influenza A/B in Point-of-Care and Non-Laboratory Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aptitude Medical Systems (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TP-23-003
Record Dates: First submitted 2023-08-25; First posted 2024-01-05 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: SARS-CoV-2 Infection; Influenza A; Influenza B
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Masking Description: Some participants will know their SOC diagnosis before completing testing on our device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- OTC Study (Experimental): This OTC study will take place in simulated home environments which will be set up within or near clinical settings (e.g., urgent care facilities). The study will enroll symptomatic subjects only. Candidate samples will be self-collected by participants (or collected by a guardian for participants under the age of 14 years) and comparator samples will be collected by a healthcare practitioner with informed consent and Institutional Review Board (IRB) approval. Each sample will be coded for confidentiality.
  Interventions: Diagnostic Test: Aptitude Medical Systems Metrix COVID/Flu Test

INTERVENTIONS:
Diagnostic Test: Aptitude Medical Systems Metrix COVID/Flu Test — The Metrix COVID/Flu Test is a real-time reverse transcription loop-mediated isothermal amplification reaction (RT-LAMP) test that has been designed to detect viral RNA from SARS-CoV-2, Influenza A, and Influenza B via electrochemical detection using the Metrix Reader. Detection of SARS-CoV-2 gene targets will produce a positive SARS-CoV-2 result, detection of the Flu A gene target will produce a positive Flu A result, and detection of the Flu B gene target will produce a positive Flu B result. If no target is detected and the internal control amplifies, the result is negative. If no amplification is detected in any of the channels, an invalid result is displayed.

SUMMARY:
The Metrix COVID/Flu Test will be evaluated for use in Point-of-Care and Non-Laboratory settings in a home testing environment utilizing the clinical study design described herein. The study will take place in simulated home environments which will be set up within or near active clinical settings (e.g., urgent care facilities). This will be a prospective study conducted at three or more investigational sites located within the United States for the clinical validation of the Metrix COVID/Flu Test for the differential detection of SARS-CoV-2, Influenza A, and Influenza B in AN swab or saliva samples. Additional sites may be added to the study in order to meet minimum subject/sample enrollment requirements and geographic prevalence of respiratory virus infections. One or more investigational sites outside of the US (at which participants are required to be fluent in English) may also be included in the study depending on enrollment needs and geographical/seasonal prevalence of respiratory virus infections. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay for the detection of SARS-CoV-2, Flu A, and/or Flu B.

DETAILED DESCRIPTION:
The Metrix COVID/Flu Test will be evaluated for OTC use in a home use testing environment utilizing the clinical study design described herein. The study will take place in simulated home environments which will be set up within or near active clinical settings (e.g., urgent care facilities). This will be a prospective study conducted at three or more investigational sites located within the United States for the clinical validation of the Metrix COVID/Flu Test for the differential detection of SARS-CoV-2, Influenza A, and Influenza B in AN swab or saliva samples. Additional sites may be added to the study in order to meet minimum subject/sample enrollment requirements and geographic prevalence of respiratory virus infections. One or more investigational sites outside of the US (at which participants are required to be fluent in English) may also be included in the study depending on enrollment needs and geographical/seasonal prevalence of respiratory virus infections. Comparator testing will be performed to determine the infection status of each sample for comparison to results generated by the candidate test. The primary comparator for the study will be an FDA-cleared assay for detection of SARS-CoV-2, Flu A, and Flu B.

The candidate device, Metrix COVID/Flu Test, will be evaluated with two specimen types - saliva and AN swab. Each Metrix COVID/Flu Test kit contains all supplies needed to test either a saliva or AN swab sample, including a corresponding QRI for each specimen type. It is possible for participants to elect to provide only a single sample type for the study; however, both sample types should be collected when possible. If participants will be testing both saliva and AN swab samples, the AN swab test should be conducted first. If participants elect to provide only a single sample type, the AN swab will be prioritized.

This OTC study will take place in simulated home environments which will be set up within or near clinical settings (e.g., urgent care facilities). The study will enroll symptomatic subjects only. Candidate samples will be self-collected by participants (or collected by a guardian for participants under the age of 14 years) and comparator samples will be collected by a healthcare practitioner with informed consent and Institutional Review Board (IRB) approval. Each sample will be coded for confidentiality.

For each participant, a comparator NP swab sample will be obtained by a healthcare practitioner after testing with the candidate device. This NP swab will be tested with the FDA-cleared SARS-CoV-2, Flu A, and Flu B assay according to the IFU and will serve as the primary comparator for both saliva and AN swab samples. An additional saliva sample will also be obtained for SARS-CoV-2 analysis via a secondary comparator method, which will be used for informational purposes only. An additional AN swab sample will be collected and stored frozen and dry for later analysis to support future research validation studies.

No results from the investigational test or comparator testing will be used for clinical diagnosis, management of study participants, or to make treatment decisions.

Test results from the Metrix COVID/Flu Test (investigational test) will be compared to the test results generated from the comparator assay.

No investigational test results will be reported to a third party or used for any treatment decisions.

Results from this study will be used in support of an Emergency Use Authorization approval from the FDA.

This work is supported by funding provided by the Biomedical Advanced Research and Development Authority (BARDA), contract number 75A50123C00013.

ELIGIBILITY:
Inclusion Criteria:

1. Participant or guardian understands and is able and willing to provide written informed consent, and assent where applicable, prior to study enrollment.
2. Male or female aged 2 years or older
3. Participant is currently exhibiting fever, or one or more symptoms associated with COVID-19 and/or influenza (such as, but not limited to, chills, cough, shortness of breath or difficulty breathing, fatigue, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting or diarrhea). Participant must still be exhibiting symptoms on the day of sample collection.
4. Participant has not eaten, consumed a beverage, smoked, brushed their teeth, gargled with mouth wash, or chewed gum for 30 minutes prior to collecting a saliva sample.
5. Participant or guardian agrees to read, and is able to read with understanding, each of the saliva and/or AN swab QRI prior to beginning the operation of each of the Metrix COVID/Flu Test.
6. Participant or guardian is able and willing to contribute the required saliva and/or swab samples for testing and understands and is able and willing to sign the study informed consent.

Exclusion Criteria:

1. Participant does not understand and/or is not able and willing to sign the study informed consent and/or assent.
2. Participant or guardian is not able to comply with saliva or nasal swab collection requirements following the QRI.
3. Participant has previously provided a sample for the study.
4. Participant has had seasonal influenza and/or the SARS-CoV-2 vaccine within the past 5 days.
5. Participant is not able to tolerate sample collection.
6. Participant is currently undergoing antiviral treatment such as baloxavir marboxil (trade name Xofluza®), oseltamivir (Tamiflu®), zanamivir (Relenza®), and peramivir (Rapivab®).
7. Participants currently undergoing treatment and/or within the past thirty (30) days with prescription medication to treat novel Coronavirus SARS-CoV-2 infection, which may include but is not limited to Remdesivir (Veklury), Paxlovid, molnupiravir or receiving convalescent plasma therapy for SARS-CoV-2.
8. Participants who have had a nasal wash or aspirate as part of their standard of care treatment on day of study visit prior to the study sample collection.
9. Participants who have had recent craniofacial injury or surgery, including to correct deviation of the nasal septum, within the previous six (6) months.
10. Participants who do not understand/read the English language.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 614 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2025-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yang, PhD, Principal Investigator — Aptitude Medical Systems
Locations (3):
- United States (3):
  - American Family Care, Trussville, Alabama
  - Central Coast Laboratories, Goleta, California
  - American Family Care, Chelmsford, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited who displayed symptoms similar to COVID and Flu infections, themselves or a guardian could understand English, and were greater than the age of 2 years old.
Pre-assignment Details: N/A, all comers approach
Period: Overall Study
Arm/Group | OTC Study
Started | 614
Completed | 556
Not Completed | 58

BASELINE CHARACTERISTICS:
Arm/Group | OTC Study
Number analyzed (Participants) | 556
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48
  Between 18 and 65 years | 473
  >=65 years | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364
  Male | 192
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Self or Assisted Testers [Count of Participants; unit: Participants] — Number of Self versus Assisted Testers
  Participants
    Self Tester | 527
    Assisted Tester | 29

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Detection of RNA From SARS-CoV-2, Influenza A, and Influenza B ; Positive Percent Agreement Performance Comparison of Candidate Device (Metrix) vs FDA-Cleared Comparator Assay
Description: Qualitative detection of RNA from SARS-CoV-2, Influenza A, and Influenza B in unprocessed saliva and/or AN swab samples. The primary objective is to evaluate the performance (positive percent agreement, negative percent agreement, and 95% confidence intervals) of the Metrix COVID/Flu Test for qualitative, differential detection of SARS-CoV-2, Influenza A, and/or Influenza B RNA using AN swab and saliva samples. Comparator testing will determine the infection status of each sample for comparison to the candidate test. The primary comparator will be an FDA-cleared assay that detects SARS-CoV-2, Flu A, and Flu B. Positive Percent Agreement (PPA) is the number of positive specimens identified by the candidate test divided by the total true positives per the comparator.
Time Frame: 45 minutes
Measure: Number (95% Confidence Interval); unit: PPA
Arm/Group | OTC Study
Number analyzed (Participants) | 556
PPA
  PPA - SARS-CoV-2 | 95.5 [88.9 to 98.2]
  PPA - Influenza A | 95.8 [88.5 to 98.6]
  PPA - Influenza B | 95.2 [84.2 to 98.7]

2. Primary Outcome: Qualitative Detection of RNA From SARS-CoV-2, Influenza A, and Influenza B ; Negative Percent AgreementPerformance Comparison of Candidate Device (Metrix) vs FDA-Cleared Comparator Assay
Description: Qualitative detection of RNA from SARS-CoV-2, Influenza A, and Influenza B in unprocessed saliva and/or AN swab samples. The primary objective is to evaluate the performance (positive percent agreement, negative percent agreement, and 95% confidence intervals) of the Metrix COVID/Flu Test for qualitative, differential detection of SARS-CoV-2, Influenza A, and/or Influenza B RNA using AN swab and saliva samples. Comparator testing will determine the infection status of each sample for comparison to the candidate test. The primary comparator will be an FDA-cleared assay that detects SARS-CoV-2, Flu A, and Flu B. Negative Percent Agreement (NPA) is the number of negative specimens identified by the candidate test divided by the total true negatives per the comparator.
Time Frame: 45 minutes
Measure: Number (95% Confidence Interval); unit: NPA
Arm/Group | OTC Study
Number analyzed (Participants) | 556
NPA
  NPA - SARS-CoV-2 | 99.6 [98.5 to 99.9]
  NPA - Influenza A | 99.4 [98.2 to 99.8]
  NPA - Influenza B | 99.4 [98.3 to 99.8]

ADVERSE EVENTS:
Time Frame: From enrollment to end of test, ~1 hour
Arm/Group | OTC Study
All-Cause Mortality (participants affected / at risk) | 0/556
Serious Adverse Events (participants affected / at risk) | 0/556
Other Adverse Events (participants affected / at risk) | 0/556

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT06191393/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT06191393/ICF_001.pdf